CLINICAL TRIAL: NCT02810782
Title: Pharmacological Treatment of Narcotic Neonatal Withdrawal
Brief Title: How to Treat Opiate Withdrawal in Neonates
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UZH-NAS01
Record Dates: First submitted 2009-06-02; First posted 2016-06-23 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2019-12

CONDITIONS: Neonatal Abstinence Syndrome
Keywords: opiate dependence; withdrawal; newborn
MeSH Terms: conditions — Neonatal Abstinence Syndrome; Opioid-Related Disorders | interventions — Phenobarbital; Chlorpromazine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Phenobarbital (Experimental): Phenobarbitone loading dose 10 mg/kg body weight maintenance dose 0.83 mg/kg body weight every 4 hours
  Interventions: Drug: Phenobarbital
- Chlorpromazine (Active Comparator): Chlorpromazine loading dose 0.5 mg/kg body weight maintenance dose 0.25 mg/kg every 4 hours
  Interventions: Drug: Chlorpromazine
- Morphine (Active Comparator): Morphine (tinctura opii) 0.25 mg/kg body weight every 4 hours
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Phenobarbital — Phenobarbital per os
  Other Names: Phenobarbitone
  Arms: Phenobarbital
Drug: Chlorpromazine — Chlorpromazine per os
  Other Names: Largactil
  Arms: Chlorpromazine
Drug: Morphine — Morphine per os
  Other Names: tinctura opii
  Arms: Morphine

SUMMARY:
Three different drugs are used in a randomised, double blind, clinical multi-centre trial with three arms. Major objective is to investigate the duration of drug treatment based on the Finnegan score. Secondary objectives are to document weight gain, the need for adding a second drug when the first drug is not effective enough and possible side effects such as convulsions.

DETAILED DESCRIPTION:
Background: Neonatal narcotic abstinence syndrome is an important medical, social and financial problem. Several drugs are used to treat the withdrawal symptoms in neonates that have been exposed to opiates in utero, but there is no consensus which one is best.

Goal: Three different drugs are used in a randomised, double blind, clinical multi-centre trial with three arms. Major objective is to investigate the duration of drug treatment based on the Finnegan score. Secondary objectives are to document weight gain, the need for adding a second drug when the first drug is not effective enough and possible side effects such as convulsions.

Methods: Neonates born after 34 completed weeks of gestation with meconium proven antenatal opiate exposure and parental informed consent are included. Infants with severe malformation are excluded. Each infant is assessed every eight hour by a modified Finnegan score. When 9 points are exceeded drug treatment is started and dose increased stepwise according to the score. The masqued solution applied orally contains morphine, phenobarbital or chlorpromazine. When the maximum dose does not reduce the score, a second randomisation and one of the two remaining drugs is added, again in a blinded way.

A total of 120 infants, 40 in each group will be included in the study.

ELIGIBILITY:
Inclusion Criteria:

* Neonates of mothers who consumed opiates during pregnancy
* Born after 34 completed weeks of pregnancy
* Parents' informed consent

Exclusion Criteria:

* Preterm birth before 34 0/7 gestational weeks
* Severe malformation
* Illness requiring respiratory assistance or catecholamines
* Negative meconium drug test

Ages: 1 Hour to 3 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2001-06; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Duration of treatment | 0 to 42 days
  Treatment is reduced stepwise until withdrawal symptoms have gone

SECONDARY OUTCOMES:
Incidence of convulsions | Whole time of hospitalisation (up to 10 weeks)
Weight gain | through study completion, up to 10 weeks
Treatment failures (need for adding second medication) | through study completion, up to 10 weeks
  Need for additional drug if investigational drug does not control withdrawal symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Hans U Bucher, Prof, Study Chair — University of Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zimmermann U, Rudin C, Duo A, Held L, Bucher HU; Swiss neonatal abstinence syndrome study group. Treatment of opioid withdrawal in neonates with morphine, phenobarbital, or chlorpromazine: a randomized double-blind trial. Eur J Pediatr. 2020 Jan;179(1):141-149. doi: 10.1007/s00431-019-03486-6. Epub 2019 Nov 6. PMID 31691849